CLINICAL TRIAL: NCT00796250
Title: Efficacy of Infliximab as "Bridging Therapy" in the Treatment of Patients Affected by Corticodependent Crohn's Disease Under Standard Treatment With Azathioprine
Brief Title: Efficacy of Infliximab in the Treatment of Patients Affected by Corticodependent Crohn's Disease (P02732)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to poor patient recruitment, a decision was made to terminate this trial.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P02732
Record Dates: First submitted 2008-11-21; First posted 2008-11-24 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Infliximab; Azathioprine; Prednisolone; prednisolone phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental)
  Interventions: Biological: Infliximab; Drug: AZA; Drug: Placebo Prednisolone
- Group B (Active Comparator)
  Interventions: Drug: Prednisolone; Drug: AZA; Biological: Placebo Infliximab

INTERVENTIONS:
Biological: Infliximab — Patients in this group were treated with azathioprine (AZA), infliximab, and placebo prednisolone. Infliximab was to be administered at a dose of 5 mg/kg at Visit 2 (Week 0), and at Weeks 2, 6, and 14 (total of four infusions). Infliximab infusions were administered by the investigators in the hospital during the patient's visit, usually in the morning.
  Other Names: Remicade; SCH 215596
  Arms: Group A
Drug: AZA — Patients in this group were treated with AZA, infliximab, and placebo prednisolone. All patients were treated with AZA, by oral use, with a 2 mgkg dose a day until the end of the study (30 weeks).
  Other Names: Imuran
  Arms: Group A
Drug: Placebo Prednisolone — Patients in this group were treated with AZA, infliximab, and placebo prednisolone. Placebo prednisolone was to be administered by oral use.
  Other Names: Placebo
  Arms: Group A
Drug: Prednisolone — Patients in this group were treated with AZA, prednisolone, and placebo infliximab. Prednisolone was to be administered by oral use, with the decreasing dose of 40 mg a day, 35 mg a day, 30 mg a day and 25 mg a day every week for each dosage, respectively; 20 mg a day for five weeks; 15 mg a day, 10 mg a day and 5 mg a day for one week for each dosage respectively, until discontinuation.
  Other Names: Pediapred
  Arms: Group B
Drug: AZA — Patients in this group were treated with AZA, prednisolone, and placebo infliximab. All patients were treated with AZA, by oral use, with a 2 mgkg dose a day until the end of the study (30 weeks).
  Other Names: Imuran
  Arms: Group B
Biological: Placebo Infliximab — Patients in this group were treated with AZA, prednisolone, and placebo infliximab. Placebo infliximab was to be administered at Visit 2 (Week 0), and at Weeks 2, 6, and 14 (total of four infusions). Infliximab infusions were administered by the investigators in the hospital during the patient's visit, usually in the morning.
  Other Names: Placebo
  Arms: Group B

SUMMARY:
This is a double-blind, double-dummy, prednisolone-controlled, multi-center, randomized, parallel-group clinical study to evaluate the therapeutic efficacy of repeated infliximab infusions in order to maintain Crohn's disease remission at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female patients with age between 18 and 65 years.
* Patients suffering from corticodependent Crohn's disease, in reheightening phase, with CDAI value >=220.
* Patients able to participate and to comply with the study.
* Patients with adequate bone marrow stock: GB >=3.5x109/L, PLTs >=100 x 103, Hb >=9 gr/dL.
* Patients able and willing to give written informed consent.

Exclusion Criteria:

* Patients with abscesses or active perianal diseases.
* Clinically symptomatic and/or with retrodilatation intestinal stenosis.
* Patients previously treated with infliximab.
* Patients with history of allergy to murine proteins.
* Treatment with immunosuppressant such as AZA, 6-mercaptopurine, methotrexate and cyclosporine A during the previous 3 months.
* Positive feces exams for intestinal pathogens, parasitic or toxin of clostridium difficilis.
* Tuberculosis (TBC) both active and inactive, evaluated by means of a detailed description (personal history of tuberculosis or possible previous contact with a source of TBC infection), and appropriate screening tests, Thorax Rx, tuberculin test.
* Presence of severe infections such as hepatitis, pneumonia, pyelonephritis within the past 3 months before the enrolment. Less severe infections, such as those in charge of the upper respiratory tract (cold syndrome), are not considered exclusion criteria as well as the uncomplicated urinary tract infections, contracted during the previous 3 months before study inclusion.
* Ongoing infections due to CMV, pneumocystis carinii, atypical mycobacterium. Proved HIV infection, presence of ARC or AIDS.
* Necessity during the study of elective or emergency surgical operation.
* Altered hepatic function: total bilirubin >=1.5 times the upper limit of the normal ranges (UNL), AST (SGOT) >=2 UNL, phosphatase alkaline >=2.5 UNL, or PTT - INR >=1.5 UNL.
* Altered renal function: creatinine >=1.5 mg.
* Presence of serious concomitant illnesses (cardiac, pulmonary, neurological diseases).
* History of pathology in charge of the haemopoietic system and of lymphoproliferative diseases such as lymphoma, lymphadenopathies of unusual localisation (i.e. at the nape, epitochlear or periaortic) or splenomegaly.
* Presence of neoplastic or pre-neoplastic lesions, or history of neoplasm in the past 5 years.
* Presence or history of drug or alcohol abuse.
* Pregnant or lactating women.
* Women of childbearing potential without adequate contraception except in case of surgical menopause. These methods of birth control should also be used during the 6 months after the last infusion.
* Contraindications for AZA (i.e. lymphoproliferative diseases, leukopenia) and prednisolone (i.e. peptic ulcer, systemic fungal infections) as laid out in the summary of product characteristics.
* Hyperamylasemia >=1.5 times the upper limit of the normal ranges.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2003-11-01 (Actual); Primary Completion 2005-01-01 (Actual); Study Completion 2005-01-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the therapeutic efficacy of repeated infliximab infusions in order to maintain Crohn's disease remission (Crohn's disease Activity Index [CDAI] <=150) at the end of the study. | Week 30

SECONDARY OUTCOMES:
Tolerability evaluation (labs parameters, vital signs, adverse events). | At each visit.
Quality of life assessment, by IBDQ questionnaire. | Baseline, Week 10, and Week 30.

REFERENCES:
- [Result] Leombruno JP, Nguyen GC, Grootendorst P, Juurlink D, Einarson T. Hospitalization and surgical rates in patients with Crohn's disease treated with infliximab: a matched analysis. Pharmacoepidemiol Drug Saf. 2011 Aug;20(8):838-48. doi: 10.1002/pds.2132. Epub 2011 Jun 17. PMID 21688345
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html